CLINICAL TRIAL: NCT04634136
Title: Full-spectrum Medical Canabis Product (HemPhar) With a CBD:THC Ratio of 10:1 for Treatment of Spasticity in Children and Young Adults With Severe Forms of Cerebral Palsy
Brief Title: Full-spectrum Medical Cannabis for Treatment of Spasticity in Patients With Severe Forms of Cerebral Palsy
Acronym: HemPhar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: PharmaHemp (Unknown); University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Principal Investigator, Damjan Osredkar, Associate Professor of Pediatrics, University Medical Centre Ljubljana
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0120-162/2017/8
Record Dates: First submitted 2020-11-04; First posted 2020-11-18 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2023-05

CONDITIONS: Children, Adult; Spastic Cerebral Palsy; Quality of Life; Cannabis; Physical Disability
Keywords: cerebral palsy; severe spasticity; child; cannabis treatment; quality of life; young adult
MeSH Terms: conditions — Cerebral Palsy; Marijuana Abuse; Muscle Spasticity | interventions — Electrocardiography; compact-colony-forming active substance

STUDY DESIGN:
Intervention Model Description: Active substance: Full-spectrum medical cannabis product of CBD/THC ratio 10:1.
  Arm 1: Active substance. The starting dose will be 0,08 mg THC per kilo body weight daily in 2 divided doses which will gradually be increased (escalating dose of 0,08 mg THC kg/d) until maximal dose of 1 mg/kg/d.
  Arm 2: Placebo
  Crossover: After 6 weeks Arm 2 will also receive the active substance and patients in both arms will continue receiving the active substance for the next 6 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo product will be of the same quantity and apperance (same packaging) as the active substance. All partricipants will be blinded to relevant patient data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Substance: Full-spectrum Medical Canabis Product (HemPhar) (Active Comparator): For research purposes the investigators will use a preparation in the form of drops, containing full-spectrum medical cannabis extract (HemPhar) with THC:CBD ratio 1:10, and other cannabinoids as well, provided by Pharmahemp, GMP-certified medical cannabis producer.
  Interventions: Diagnostic Test: Lab tests; Diagnostic Test: ECG; Diagnostic Test: Cannabinoid Levels; Drug: Full-spectrum Medical Canabis Product (HemPhar); Diagnostic Test: Spasticity level according to modified Ashworth scale (Bohannon); Diagnostic Test: Gross Motor Function Measure; Diagnostic Test: Borg rating of perceived exertion scale; Diagnostic Test: Edmonton symptom assessment system
- Placebo (Placebo Comparator): For research purposes the investigators will use a placebo in the form of drops, containing oil only, provided by Pharmahemp, GMP-certified medical cannabis producer.
  Interventions: Diagnostic Test: Lab tests; Diagnostic Test: ECG; Drug: Placebo; Diagnostic Test: Spasticity level according to modified Ashworth scale (Bohannon); Diagnostic Test: Gross Motor Function Measure; Diagnostic Test: Borg rating of perceived exertion scale; Diagnostic Test: Edmonton symptom assessment system

INTERVENTIONS:
Diagnostic Test: Lab tests — CBC and differential counts, blood electrolytes, magnesium, calcium, phosphorus, urea & creatinine, liver enzymes (AST, ALT, gGT)
  Other Names: Basic hematology and biochemistry
Diagnostic Test: ECG — Electrocardiogram
Diagnostic Test: Cannabinoid Levels — Determination of levels of cannabidiol (CBD) and delta-9-tetrahydrocannbinol (THC) for determination of levels at following time(s) after ingestion: 0, 1, 2, 4, 8 and 24 hours.
  Other Names: Pharmacokinetics of cannabinoids
  Arms: Active Substance: Full-spectrum Medical Canabis Product (HemPhar)
Drug: Full-spectrum Medical Canabis Product (HemPhar) — Active substance
  Other Names: Active substance
  Arms: Active Substance: Full-spectrum Medical Canabis Product (HemPhar)
Drug: Placebo — Placebo
  Arms: Placebo
Diagnostic Test: Spasticity level according to modified Ashworth scale (Bohannon) — A trained physiotherapist will assess spasticity level according to modified Ashworth scale (Bohannon), which is 6-level scale for assessment of spasticity.
  Modified Ashworth/Bohannon Scoring Scale (Bohannon and Smith, 1987):
  0 No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+ Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of movement (ROM )
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
  Best score is 0 (no spasticity), worst score is 4 (severe spasticity).
Diagnostic Test: Gross Motor Function Measure — A trained physiotherapist will assess Gross Motor Function Measure (GMFM-88) which is commonly used in the evaluation of gross motor function in children with cerebral palsy
  The Gross Motor Function Measure-88 (GMFM-88) is a standardized observational instrument developed to measure change in gross motor function over time. The test consists of 88 items categorized in five dimensions (Dimension A: lying and rolling, Dimension B: sitting, Dimension C: crawling and kneeling, Dimension D: standing and Dimension E: walking, running and jumping). The test was conducted as described in the GMFM-88 manual . A percentage score as compared to maximum is calculated for each dimension and for the total score of the five dimensions.
  Reference curves exist for GMFM-88 for each age group.
  Floor score is 4 (minimum score / worst), ceiling score (maximum score / best) is 75.
Diagnostic Test: Borg rating of perceived exertion scale — Borg rating of perceived exertion scale
Diagnostic Test: Edmonton symptom assessment system — Edmonton symptom assessment system and general impression scale (1 - very much improved; 7 - very much worse).

SUMMARY:
The proposed study is a double-blind, placebo-controlled, cross over study on 60 children aged 5 to 25 years with severe spasticity related to cerebral palsy (CP), level IV and V with full-spectrum medical cannabis product of CBD/THC ratio 10:1.

DETAILED DESCRIPTION:
Test components:

A) Active: Full-spectrum medical cannabis with ratio of CBD:THC 10:1 (HemPhar)

B) Placebo (both of the same producer)

Study Steps

1. Informed consent should be signed by parents/caregivers.
2. Weight of the participant should be determined and an IV line inserted. The following lab tests should be performed: CBC and differential counts, blood electrolytes, magnesium, calcium, phosphorus, urea & creatinine, liver enzymes (AST, ALT, gGT)
3. ECG performed and analyzed
4. A trained physiotherapist will perform the following motor assessments: spasticity level according to modified Ashworth scale (Bohannon), function/activity assessment with the use of Gross Motor Function Measure scale (GMFM-88) and assessment of muscle power with dynamometer.
5. Randomization of patients into one of the two arms of the study
6. Active substance or placebo are introduced thereafter (as an oral oily solution for oral application) in a starting dose of 0.08 mg/kg body weight (BWt)/day divided in 2 doses (the dose is according to the THC content). The dose is gradually increased, every 3 days for 0.08 mg THC/ kg BWt/day, until the maximum dose of 1 mg THC/kg BWt/day is reached, or else until adverse effects are noted. It is expected that the average dose will be 0.33 mg/kg BWt per day.
7. The parents/caregivers are given questionnaires/scales and also given oral instructions on how to fulfil them (Edmonton scale, Borg scale and Global Impression of Change - GIC) and the paper to take down notes on possible side/adverse effects while taking the preparation (either active substance or placebo).
8. After 6 weeks of taking the substance or at the premature end of the study again the lab tests will be performed as well as the motor assessment by the physiotherapist (as above at inclusion).
9. In patients, who have been receiving placebo for the first 6 weeks, the active substance is given for the next 6 weeks, as described above (under 6). The patients who have been receiving the active substance for the first 6 weeks will continue to do so for the next 6 weeks.
10. Additional blood samples are taken at 6 weeks in both groups for analysis of levels of cannabidiol (CBD) as well as delta-9-tetrahydrocannbinol (THC) - around 4 ml of blood for determination of both levels at time(s) after ingestion: 0, 1, 2, 4, 8 and 24 hours.
11. At the end of the study (after 12 weeks) again repeat:

    1. CBC and differential counts, blood electrolytes, magnesium, calcium, phosphorus, urea & creatinine, liver enzymes (AST, ALT, gGT)
    2. ECG
    3. Motor assessments by a physiotherapist (Ashworth/Bohannon, GMFM 88, dynamometer)
    4. Pharmacokinetics: 4 ml of blood for determination of phamacokinetics after ingestion of the last dose (as in point 10 above)
12. Evaluation of the questionnaires

NOTE: if severe side/adverse effects are noted, the test compound should be stopped immediately. If mild/moderate side/adverse effects are noted, the test component should be gradually stopped: for 0,08 mg/kg BWt/day, every 3 days.

ELIGIBILITY:
Inclusion criteria:

* With confirmed diagnosis of cerebral palsy (CP) and classified according to the Gross Motor Function Classification System (GMFCS) as level IV or V
* With spastic unilateral or spastic bilateral type of CP
* Those children/young adults whose parents/caregivers were informed about the aims of the study and have signed the Informed consent form

Exclusion criteria:

* Other proven diseases/conditions with the prevalence of spastic type of muscle tone (e.g. neurodegenerative, metabolic, etc.), and children with liver disease
* Other forms of CP (dyskinetic, ataxic)
* History of psychiatric illness/condition in the family

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Effect on spasticity (6w; FSMC vs placebo) | 6 weeks
  A trained physiotherapist will assess spasticity level according to modified Ashworth scale (Bohannon), which is 6-level scale for assessment of spasticity.
  Modified Ashworth/Bohannon Scoring Scale (Bohannon and Smith, 1987):
  0 No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+ Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of movement (ROM )
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
  Best score is 0 (no spasticity), worst score is 4 (severe spasticity).
Effect on Gross Motor Function Measure (6w; FSMC vs placebo) | 6 weeks
  A trained physiotherapist will assess Gross Motor Function Measure (GMFM-88) which is commonly used in the evaluation of gross motor function in children with cerebral palsy
  The Gross Motor Function Measure-88 (GMFM-88) is a standardized observational instrument developed to measure change in gross motor function over time. The test consists of 88 items categorized in five dimensions (Dimension A: lying and rolling, Dimension B: sitting, Dimension C: crawling and kneeling, Dimension D: standing and Dimension E: walking, running and jumping). The test was conducted as described in the GMFM-88 manual . A percentage score as compared to maximum is calculated for each dimension and for the total score of the five dimensions.
  Reference curves exist for GMFM-88 for each age group.
  Floor score is 4 (minimum score / worst), ceiling score (maximum score / best) is 75.
Effect on spasticity (12w; 12w-FSMC vs 6w-FSMC) | 12 weeks
  A trained physiotherapist will assess spasticity level according to modified Ashworth scale (Bohannon), which is 6-level scale for assessment of spasticity
  Modified Ashworth/Bohannon Scoring Scale (Bohannon and Smith, 1987):
  0 No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+ Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of movement (ROM )
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
  Best score is 0 (no spasticity), worst score is 4 (severe spasticity).
Effect on Gross Motor Function Measure (12w; 12w-FSMC vs 6w-FSMC) | 12 weeks
  A trained physiotherapist will assess Gross Motor Function Measure (GMFM-88) which is commonly used in the evaluation of gross motor function in children with cerebral palsy.
  The Gross Motor Function Measure-88 (GMFM-88) is a standardized observational instrument developed to measure change in gross motor function over time. The test consists of 88 items categorized in five dimensions (Dimension A: lying and rolling, Dimension B: sitting, Dimension C: crawling and kneeling, Dimension D: standing and Dimension E: walking, running and jumping). The test was conducted as described in the GMFM-88 manual . A percentage score as compared to maximum is calculated for each dimension and for the total score of the five dimensions.
  Reference curves exist for GMFM-88 for each age group.
  Floor score is 4 (minimum score / worst), ceiling score (maximum score / best) is 75.
Safety and tolerability of FSMC | 12 weeks
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]

CONTACTS AND LOCATIONS:
Overall Officials: Damjan Osredkar, MD, PhD, Study Director — UMC Ljubljana
Locations (2):
- Slovenia (2):
  - PharmaHemp, Ljubljana
  - University Medical Centre Ljubljana, Ljubljana